CLINICAL TRIAL: NCT05075980
Title: HEADLIGHT: Hypofractionated Proton Therapy for Head and Neck Cancers
Brief Title: Intensity Modulated Proton or X-Ray Therapy After Surgery for Treatment of Head and Neck Cancer, the HEADLIGHT Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2171; NCI-2021-09706 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-000973 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Carcinoma; Head and Neck Carcinoma of Unknown Primary; Hypopharyngeal Carcinoma; Laryngeal Carcinoma; Metastatic Malignant Neoplasm in the Lymph Nodes; Nasal Cavity Carcinoma; Oral Cavity Carcinoma; Oropharyngeal Carcinoma; Paranasal Sinus Carcinoma; Salivary Gland Carcinoma; Cutaneous Squamous Cell Carcinoma of the Head and Neck; Locally Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Lymphatic Metastasis; Mouth Neoplasms; Oropharyngeal Neoplasms; Paranasal Sinus Neoplasms; Salivary Gland Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Magnetic Resonance Spectroscopy; X-Rays; Specimen Handling; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm A (IMPT, IMRT, cisplatin) (Experimental): Patients undergo IMPT or IMRT for 18 sessions over 24 days in the absence of disease progression or unacceptable toxicity. Patients may receive cisplatin IV over 1-2 hours per standard of care. Patients undergo CT or MRI and PET/CT or PET/MRI during screening and follow-up. Patients may also undergo blood sample collection throughout the trial.
  Interventions: Drug: Cisplatin; Procedure: Intensity-Modulated Proton Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection; Radiation: Intensity-Modulated Radiation Therapy
- Arm B (IMPT, cisplatin) (Experimental): Patients undergo IMPT for 15 sessions over 19 days in the absence of disease progression or unacceptable toxicity. Patients may receive cisplatin IV over 1-2 hours per standard of care. Patients undergo CT or MRI and PET/CT or PET/MRI during screening and follow-up. Patients may also undergo blood sample collection throughout the trial.
  Interventions: Drug: Cisplatin; Procedure: Intensity-Modulated Proton Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection
- Arm C (IMRT, cisplatin) (Experimental): Patients undergo IMRT for 15 sessions over 19 days in the absence of disease progression or unacceptable toxicity. Patients may receive cisplatin IV over 1-2 hours per standard of care. Patients undergo CT or MRI and PET/CT or PET/MRI during screening and follow-up. Patients may also undergo blood sample collection throughout the trial.
  Interventions: Drug: Cisplatin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection; Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Intensity-Modulated Proton Therapy — Undergo IMPT
  Other Names: IMPT
  Arms: Arm A (IMPT, IMRT, cisplatin); Arm B (IMPT, cisplatin)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI or PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Specimen Collection
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Intensity Modulated X-ray Therapy
  Arms: Arm A (IMPT, IMRT, cisplatin); Arm C (IMRT, cisplatin)

SUMMARY:
This clinical trial studies how well intensity modulated proton therapy (IMPT) or intensity modulated X-ray (radiation) therapy (IMRT) works after surgery in treating patients with head and neck cancer. IMPT is a type of radiation therapy that allows for the most accurate application of proton radiation to the tumor and has the potential to reduce treatment-related side effects. IMRT is a type of 3-dimensional radiation therapy that uses computer-generated images to show the size and shape of the tumor. Thin beams of x-ray radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor. IMPT may work as well as IMRT after surgery in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the local-regional control among subjects in each arm at 2 years after study registration.

II. To evaluate difference in MD Anderson Dysphagia Inventory (MDADI) score between patients with proton and intensity-modulated radiation therapy (IMRT) adjuvant radiation.

SECONDARY OBJECTIVES:

I. To determine overall survival, progression free survival, local, regional, distant recurrence risks, and infield and outfield recurrence in the trial at 2 years after study registration.

II. To determine the rate of grade 3+ acute adverse events (from treatment start to 30 days after radiation completion date).

III. To determine the rate and severity of late solicited toxicities. IV. To determine the incidence of secondary acute effects attributable to radiotherapy (e.g., percutaneous endoscopic gastrostomy [PEG] tube placement, duration and dose of narcotic analgesia required, weight loss, and hospitalization days).

V. To determine the impact of treatment on patient-reported quality of life. VI. To objectively quantify the severity of oral mucositis during and following radiotherapy.

EXPLORATORY OBJECTIVES:

I. To estimate direct and indirect costs of the study regimen and compare these with standard of care treatment techniques.

II. To correlate histopathologic, molecular, and tumor genetic/epigenetic alterations with clinical outcomes.

III. To correlate circulating biomarkers (micro ribonucleic acid [miRNA], circulating tumor deoxyribonucleic acid [ctDNA]) with clinical outcomes.

IV. To determine adverse events and patient reported outcomes related to abbreviated concomitant chemotherapy.

V. To qualitatively evaluate patient beliefs regarding tradeoffs of cancer control, treatment time, cost, acute side effects, and late side effects.

VI. To determine cancer outcomes, adverse events, and patient reported outcomes and compare across head and neck subsites, between those aged ≥ 65 to those age < 65 at date of enrollment, between male and female, and in the adjuvant population between time to total package completion (< 9 weeks vs ≥ weeks, surgery = day 0), and by treatment with and without chemotherapy.

VII. To evaluate the predictive relationship of linear energy transfer (LET) weighted modeling using an relative biologic enhancement (RBE)-based model and RBE-independent model with grade 3+ acute and late toxicity.

OUTLINE: Patients who already underwent surgical resection are assigned to Arm A. Patients who have undergone upfront surgical resection and need postoperative radiotherapy are assigned to Arm B or Arm C.

ARM A: Patients undergo intensity modulated proton therapy (IMPT) or IMRT for 18 sessions over 24 days in the absence of disease progression or unacceptable toxicity. Patients may receive cisplatin intravenously (IV) over 1-2 hours per standard of care. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) and positron emission tomography (PET)/CT or PET/MRI during screening and follow-up. Patients may also undergo blood sample collection throughout the trial.

ARM B: Patients undergo IMPT for 15 sessions over 19 days in the absence of disease progression or unacceptable toxicity. Patients may receive cisplatin IV over 1-2 hours per standard of care. Patients undergo CT or MRI and PET/CT or PET/MRI during screening and follow-up. Patients may also undergo blood sample collection throughout the trial.

ARM C: Patients undergo IMRT for 15 sessions over 19 days in the absence of disease progression or unacceptable toxicity. Patients may receive cisplatin IV over 1-2 hours per standard of care. Patients undergo CT or MRI and PET/CT or PET/MRI during screening and follow-up. Patients may also undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up within 21 days and then at months 3, 6, 9, 12, 15, 18, 24, 35, 48, and 60.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of a newly diagnosed non-human papillomavirus (HPV) associated malignant epithelial cancer in the head and/or neck. Diagnosis requires confirmation of p16 and/or HPV DNA negativity for oropharyngeal and unknown primary sites. p16 positivity in skin cancers is allowed
* Primary lesion located in the nasal cavity, paranasal sinuses, oral cavity, oropharynx, larynx, hypopharynx, salivary glands, lymph nodes (unknown primary or metastasis from head and neck [HN]-skin primary) or skin cancer where lymph node radiation is recommended

  * NOTE: Patients with primary lesions in the larynx must have a T3 primary, bulky T2 primary (> 6 cc), and/or at least 1 regional lymph node
* Confirmation of American Joint Committee on Cancer (AJCC) 8th edition defined M0 established by positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status (0-1 prior to initial treatment)
* Able to provide written informed consent
* Able to complete questionnaires independently or with assistance
* Willing to return to enrolling institution for follow up during the observation phase

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 2 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix and prostate cancer with a Gleason score of 6 or less
  * NOTE: If there is a history or prior malignancy, they must not be receiving ongoing anticancer treatment
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Prior radiation therapy that would have a clinically significant overlap with the intended head/neck radiation
* For Arms A and B only: Unable to receive proton therapy because of extensive metallic hardware in close proximity to treatment site, logistical circumstances, or any other reason
* Any of the following diagnoses: HPV-associated squamous cell carcinoma, germ cell tumors, hematologic malignancies, neuroendocrine malignancies, adenoid cystic carcinoma, sarcomas of bone, benign tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2035-11-15 (Estimated)

PRIMARY OUTCOMES:
Rate of local/regional control (LRF) | At 2 years
  The 2-year LRF rate will be estimated by counting the number of patients with a local or regional failure and dividing by the total number of eligible patients.

SECONDARY OUTCOMES:
Incidence of acute adverse events | Up to 3 months after radiation therapy
  The maximum grade for each type of acute adverse event will be recorded for each patient. Data will be summarized as frequencies and relative frequencies. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Incidence of late adverse events | Up to 3 years after completion of radiation therapy
  The maximum grade for each type of late adverse event will be recorded for each patient. Data will be summarized as frequencies and relative frequencies. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Incidence of secondary acute effects attributable to radiation therapy | Up to 3 months after completion of radiation therapy
  The electronic health record will be reviewed for treatments related to secondary acute effects such as PEG tube placement, duration and dose of narcotic analgesia required, weight loss, and hospitalization days.
Quality of life (QOL) and financial burden - MDADI | Up to 10 years
  MD Anderson Dysphagia Inventory (MDADI) will be utilized to assess patient reported quality-of-life and financial burden. Changes from baseline to end of therapy as well as repeated measures mixed models will be utilized to assess effect of treatment. The QOL measurements will be summarized at each time point as mean +/- standard deviation and median (minimum value, maximum value). Changes in the QOL measurements from baseline will be determined at each follow-up measurement. These will be displayed as spaghetti plots. The assessment of the changes at each time point will be done with a paired t-test or Wilcoxon signed rank test, whichever is appropriate. Scale of 0 being least and 10 being greatest effect.
Quality of life (QOL) and financial burden - EQ-5D-5L | Up to 10 years
  European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L) will be utilized to assess patient reported quality-of-life and financial burden. Changes from baseline to end of therapy as well as repeated measures mixed models will be utilized to assess effect of treatment. The QOL measurements will be summarized at each time point as mean +/- standard deviation and median (minimum value, maximum value). Changes in the QOL measurements from baseline will be determined at each follow-up measurement. These will be displayed as spaghetti plots. The assessment of the changes at each time point will be done with a paired t-test or Wilcoxon signed rank test, whichever is appropriate. Scale of 0 being least and 10 being greatest effect.
Quality of life (QOL) and financial burden - OMWQ-HN | Up to 10 years
  Oral Mucositis Weekly Questionnaire (OMWQ-HN) will be utilized to assess patient reported quality-of-life and financial burden. Changes from baseline to end of therapy as well as repeated measures mixed models will be utilized to assess effect of treatment. The QOL measurements will be summarized at each time point as mean +/- standard deviation and median (minimum value, maximum value). Changes in the QOL measurements from baseline will be determined at each follow-up measurement. These will be displayed as spaghetti plots. The assessment of the changes at each time point will be done with a paired t-test or Wilcoxon signed rank test, whichever is appropriate. Scale of 0 being least and 10 being greatest effect.
Regional recurrence rates | Up to 10 years
  The regional head and neck cancer recurrence cumulative incidence will be estimated using a competing risks method (Gooley et al.). The competing risks will be local/distant head and neck cancer recurrence and death.
Local recurrence incidence | Up to 10 years
  The local head and neck cancer recurrence cumulative incidence will be estimated using a competing risks method (Gooley et al.). The competing risks will be regional/distant head and neck cancer recurrence and death.
Distant recurrence rates | Up to 10 years
  The distant head and neck cancer recurrence cumulative incidence will be estimated using a competing risks method (Gooley et al.). The competing risks will be local/regional head and neck cancer recurrence and death.
Invasive disease-free survival (DFS) | From registration until the time of disease recurrence or death due to any cause, assessed up to 10 years
  The DFS will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% confidence intervals.
Overall survival (OS) | From registration to death due to any cause, assessed up to 10 years
  The OS will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Scott C. Lester, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (9):
- United States (9):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System - Mankato, Mankato, Minnesota
  - Mayo Clinic Radiation Therapy - Northfield, Northfield, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials